#### Cover Page for Clinical Trials Document posting

Official Title: S1400K, "A Phase II Study of ABBV-399 (Process II) in Patients with c-Met Positive Stage

IV or Recurrent Squamous Cell Lung Cancer (Lung-MAP Sub-Study)"

NCT Number: 03574753

Version Date: 10/21/20

Description:

**S1400** [NCT 02154490] is the parent study to **S1400K** [NCT 03574753].

The **<u>\$1400</u>** Lung-MAP study is considered one study under one IND consisting of:

S1400 Version Control Protocol

• S1400 Main Screening Protocol Component

Multiple Sub-Studies (or sub-protocols) Components

Each component is contained in its own separate document.

<u>S1400K</u> is one of these components. Each "component" consists of the protocol document and its associated informed consent document(s). Since each screening and sub-study component operates independently from the other components contained in Lung-MAP, each has its own version date and NCT number. This is due to the complexity of the study and how it must be entered into different computer programs.

S1400K Treatment Consent Page 1 Version Date 10/21/20

# Study Title for Study Participants: Targeted Treatment for Advanced Squamous Cell Lung Cancer

## Official Study Title for Internet Search on

http://www.ClinicalTrials.gov:

<u>S1400</u>, "A Biomarker-Driven Master Protocol for Previously Treated Squamous Cell Lung Cancer"

S1400K, "A Phase II Study of ABBV-399 (Process II) in Patients with c-Met Positive Stage IV or Recurrent Squamous Cell Lung Cancer (Lung-MAP Sub-Study)"

## What is the usual approach to my lung cancer?

Squamous cell lung cancers make up about one-fourth of non-small cell lung cancer. Various chemotherapy drugs have been shown to improve survival for patients with advanced squamous cell lung cancer. Most patients, for example, will be treated at first with a platinum-based chemotherapy (like cisplatin or carboplatin) in combination with a second chemotherapy drug such as gemcitabine, paclitaxel, docetaxel, or vinorelbine.

In addition, immunotherapy has been FDA approved for patients whose disease has gotten worse. The approval was based on results of clinical trials where patients had improved overall survival with immunotherapy compared to standard chemotherapy.

- For patients with previously untreated squamous cell lung cancer, immunotherapy options include pembrolizumab alone for tumors that have a high expression of a marker called PD-L1.
- For patients whose disease has gotten worse while receiving platinum-based chemotherapy (like cisplatin or carboplatin), immunotherapy options include pembrolizumab alone for tumors with a low tumor expression of PD-L1.
- Other available immunotherapy options are nivolumab and atezolizumab, which do not need PD-L1 expression testing.

## What are my other choices if I do not take part in this study?

Your other choices may include:

- You may choose to have the usual approach described above
- You may choose to take part in a different study, if one is available
- You may choose to get comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.



## Why is this study being done?

There are several investigational treatments that are being tested in various sub-studies as part of this study. You will have already received the information on your biomarker testing. You have been assigned to this treatment study because your tumor sample is c-MET positive. C-MET is a protein that is involved in tumor growth and exists on the surface of lung cancer cells. For this sub-study, you will be assigned to treatment with a drug called ABBV-399 (Process II). ABBV-399 (Process II) is considered investigational, which means that it has not been approved by the U.S. Food and Drug Administration (FDA). ABBV-399 (Process II) is a type of drug called an antibody-drug conjugate (ADC). ADC's are designed to more precisely deliver chemotherapy to cancer cells and spare healthy cells. ABBV-399 (Process II) binds to the protein c-MET that is expressed on the surface of lung cancer cells. After binding, the ADC enters the cell and separates the chemotherapy from the antibody so that it becomes active. The purpose of this substudy is to test the safety of ABBV-399 (Process II) and find out what effects, if any, ABBV-399 (Process II) has on people and their lung cancer. ABBV-399 (Process II) may or may not shrink your cancer and it could also cause side effects.

There will be about 44 patients taking part in this sub-study.

#### What are the study groups?

You have been assigned to this sub-study because your tumor sample is c-MET positive.

All patients will receive the study drug ABBV-399 (Process II). The study drug will be given through a vein in your body over about 30 minutes on Day 1 of every 21-day cycle.

The treatment on this study is described in the table below:

| Drug | How often is it given? | How is it given? | What days is it given on? | How long is the cycle? |
|---|---|---|---|---|
| ABBV-399<br>(Process II) | Once per cycle every 21 days | Into a vein | Day 1 | 21 days |



Another way to find out what may happen to you during the study is to read the chart below. Start reading at the top of the chart and read down, following the arrows.



## How long will I be in this study?

You will receive treatment until your disease worsens, you experience a severe side effect, or your doctor thinks you should stop taking the study treatment. After you are finished taking study treatment, the study doctor will continue to watch you for side effects and follow your condition for up to three years from the time you started treatment. At the follow up visits you will have a physical exam, blood tests, and scans. Your doctor may give you other tests or procedures if they think they are needed for the regular care of your disease.

Should your disease worsen, you have the option to participate in a different sub-study. As before, the new sub-study that you will be offered will depend on a combination of the results of the previous testing done on your tumor sample and the sub-studies available. If the tests show that your tumor has more than one biomarker that qualifies you for a different sub-study, you will be assigned to one of these sub-studies randomly (by chance). A sub-study may be available if your tumor does not have any additional biomarkers being tested or you were not eligible to participate in other sub-studies.

## What extra tests and procedures will I have if I take part in this study?

Most of the exams, tests, and procedures you will have are part of the usual approach for your cancer. However, there are some extra exams, tests, and/or procedures that you will need to have if you take part in this study.

The left-over tumor sample from your screening biomarker testing will have additional laboratory tests. The samples will be kept until there are no additional sub-studies for you to enroll in or they are used up, whichever happens first. If any tumor is left over after the laboratory studies and there are no additional sub-studies for you to enroll in, and if you agreed, it will be stored for biobanking. This was discussed in the screening consent section on optional studies.



If the exams, tests, and procedures show that you are eligible to take part in the study, and you choose to take part, then you will need the following extra tests. They are not part of the usual approach for your type of cancer.

Before you begin the study:

- o Brain CT or MRI (to check if your cancer may have spread to your brain)
- o Blood tests to assess your liver functions (GGT), kidney functions (phosphate and magnesium), and testosterone levels in men

#### During the study:

- o Brain CT or MRI (to check if your cancer may have spread to your brain)
- o Blood tests to assess your liver functions (GGT), kidney functions (phosphate and magnesium), and testosterone levels in men
- o Blood tests for studies of drug levels

Neither you nor your health care plan/insurance carrier will be billed for the following tests obtained for the purpose of this study.

- o Blood tests for studies of drug levels
- o Blood tests to assess your liver functions (GGT) kidney functions (phosphate and magnesium), and testosterone levels in men

You might receive a CT or MRI even if you were not on the study as part of your usual cancer care. You will have a CT or MRI done before you begin the study and then approximately every six weeks for the first year then every 3 months until your disease worsens and stop treatment. Your doctor will review the CT scans or other radiographic scans done to check on your tumors on a regular basis. These scans will also be sent to a central location for review. This central review is part of a total study analysis only. Information on your scans from the central review will not be sent back to you or your doctor.

The blood test to assess your liver and kidney functions and testosterone levels (males) will be done before you begin the study and at each cycle. Additional blood samples are also required for you to take part in this study.

Researchers for this study are interested in testing what happens to the study drug once it gets in your body- this is called pharmacokinetic testing. The samples will be collected on Day 1 of Cycles 1, 2, 3, and 4. One sample will be collected 30 minutes before you start treatment and another sample will be collected about an hour after treatment. At each time point you will have a single needle stick and about 1 tablespoon of blood will be collected.



## What possible risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that you may:

- Lose time at work or home and spend more time in the hospital or doctor's office than usual
- Be asked sensitive or private questions which you normally do not discuss

The treatment used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood and will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects.

Here are important points about side effects:

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.
- Some side effects may interfere with your ability to have children.
- Some side effects may be serious and may even result in death.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drug to try to reduce side effects.

Your drug medication list will be reviewed at each visit. You will be given a handout and wallet card about potential drug interactions. Your study doctor will discuss with you of any potential drug interactions.

The tables provided below show the most common and the most serious side effects that researchers know about related to ABBV-399 (Process II). There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.



#### Possible Side Effects of ABBV-399 (Process II)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving ABBV-399 (Process II), more than 20 and up to 100 may have:

- Constipation
- Nausea
- Tiredness
- Swelling of arms, legs

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving ABBV-399 (Process II), from 4 to 20 may have:

- Anemia which may cause tiredness, or may require blood transfusion
- Infection, especially when white blood cell count is low
- Diarrhea
- Vomiting
- Loss of appetite
- Pain in joints
- Numbness, tingling or pain of the hands, arms, feet and legs
- Low blood pressure which may cause feeling faint

#### RARE, AND SERIOUS

In 100 people receiving ABBV-399 (Process II), 3 or fewer may have:

- Muscle weakness
- Swelling in testis (males)

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

Reproductive risks: You should not get pregnant, breastfeed, or father a baby while in this study as the drugs used in this study could be very damaging to an unborn or newborn baby. There may be some risks that researchers do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and for 6 months after you have completed the study.

Pneumonitis, a lung inflammation not due to an infection, is a known risk of cancer therapies you may have received. Therapies such as: immunotherapy, kinase inhibitors, and a drug called ADCETRIS®. ADCETRIS® is similar to ABBV-399. It is not clear if ABBV-399 causes pneumonitis; however, pneumonitis (including some cases that have resulted in death), has been reported in patients receiving ABBV-399 in clinical trials. Your doctor may decide to delay, withhold, or discontinue ABBV-399 treatment if you and your doctor think it would be in your best interest.



#### What possible benefits can I expect from taking part in this study?

It is not possible to know at this time if the study drug/study approach is better than the usual approach, so this study may or may not help you. This study will help researchers learn things that will help people in the future.

#### Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. If you stop, you can decide whether or not to let the study doctor continue to provide your medical information to the organization running the study.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and the study is no longer in your best interest
- If new information becomes available
- If you do not follow the study rules
- If the study is stopped by the sponsor, IRB or FDA.

## What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

| For questions about your rights while in this study, call the | |
|---|---|
| (insert name of center) Institutional Review Board at | (insert telephone |
| number). (Note to Local Investigator: Contact information for patient represen | tatives or other |
| individuals at a local institution who are not on the IRB or research team but to | ake calls |
| regarding clinical trial questions can also be listed here.) | |

## What are the costs of taking part in this study?

ABBV-399 (Process II) will be supplied at no charge while you take part in this study. The cost of getting ABBV-399 (Process II) ready and giving it to you is not paid by the study sponsor so you or your insurance company may have to pay for this. It is possible that ABBV-399 (Process II) may not continue to be supplied while you are on the study. Although not likely, if this occurs, your study doctor will talk to you about your options.

You and/or your health plan/insurance company will need to pay for all of the other costs of treating your cancer while in this study, including the cost of tests, procedures, or medicines to manage any side effects, unless you are told that certain tests are supplied at no charge. Before you decide to be in the study, you should check with your health plan or insurance company to find out exactly what they will pay for.

You will not be paid for taking part in this study.



## What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a study.

#### Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The study sponsor, SWOG, and the drug company supporting the treatment sub-study you are on.
- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study.
- The Food and Drug Administration (FDA) and the National Cancer Institute (NCI) in the U.S., and similar ones if other countries are involved in the study.
- TRIAD-Your medical images with clinical study data (e.g., the treatment Group you are assigned to, etc.) will be transferred to the Ohio State University in Columbus, Ohio. Your medical images will be reviewed by physicians at this organization as part of the study analysis for this trial.
- In addition, information gained from this study may be used in the future for additional research and only that data would be provided to other scientist for future research. Your name, and any other information that could be used to identify you personally, will not be included.

## Where can I get more information?

You may visit the NCI Web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).



A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

[Note to Informed Consent Authors: The above paragraph complies with the new FDA regulation found at 21CFR50.25 (c) and must be included verbatim in all informed consent documents. The text in this paragraph cannot be revised.]

## Who can answer my questions about this study?

| You can talk to the study doctor a | about any questions or concerns you | have about this study or to |
|---|---|---|
| report side effects or injuries. Con | ntact the study doctor | (insert name of |
| study doctor[s]) at | (insert telephone number). | |

#### This section is about optional studies you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. You will not get health benefits from any of these studies. The researchers leading this optional study hope the results will help other people with cancer in the future.

The results will not be added to your medical records, nor will you or your study doctor know the results.

You will not be billed for these optional studies. You can still take part in the main study even if you say 'no' to any or all of these studies. If you sign up for but cannot complete any of the studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for each of the following studies.

## 1. Optional Additional Biopsy and Optional Sample Collections for Laboratory Studies and/or Biobanking for Possible Future Studies

Researchers are trying to learn more about cancer, diabetes, and other health problems. Much of this research is done using samples from your tissue, blood, urine, or other fluids. Through these studies, researchers hope to find new ways to prevent, detect, treat, or cure health problems.

Some of these studies may be about genes. Genes carry information about features that are found in you and in people who are related to you. Researchers are interested in the way that genes affect how your body responds to treatment.

If you choose to take part in this part of the study, the researchers would also like to ask your permission to store and use your samples and health information for medical research. The research that may be done is unknown at this time. Storing samples for future studies is called



"biobanking". The Biobank is being run by SWOG and supported by the National Cancer Institute.

#### WHAT IS INVOLVED?

If you agree to take part, here is what will happen next:

- Your specimens may be stored in the Biobank, along with samples from other people who take part. These specimens may include:
  - About 2 tablespoons of blood will be collected from a vein in your arm (at the same time as other study blood tests) on Baseline, weeks 4, 7, 10, and again if your cancer gets worse.
    - The most common risks related to drawing blood from your arm are brief pain and possibly a bruise.
  - A sample of tissue will be collected from an optional extra biopsy if your cancer gets worse after treatment on this study. Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, pain and bruising at the biopsy site, which can be treated with regular pain medications.
    - Rarely, an infection can occur. Rarely, patients may experience partial lung collapse that may require a chest tube or breathing machine. You will sign a separate consent form before the biopsy is taken. This will be a standard surgical consent form from the institution where the biopsy procedure takes place. The samples may be used to test for genes (DNA, RNA), protein or metabolites and will be kept until they are used up.
- Qualified researchers can submit a request to use the materials stored in the Biobanks. A science committee at the clinical trials organization, and/or the National Cancer Institute, will review each request. There will also be an ethics review to ensure that the request is necessary and proper. Researchers will not be given your name or any other information that could directly identify you.
- 3) Neither you nor your study doctor will be notified when research will be conducted or given reports or other information about any research that is done using your samples.
- 4) Some of your genetic and health information may be placed in central databases that may be public, along with information from many other people. Information that could directly identify you will not be included.

#### WHAT ARE THE POSSIBLE RISKS?

- 1) There is a risk that someone could get access to the personal information in your medical records or other information researchers have stored about you.
- There is a risk that someone could trace the information in a central database back to you. Even without your name or other identifiers, your genetic information is unique to you. The researchers believe the chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information.



In some cases, this information could be used to make it harder for you to get or keep a job or insurance. There are laws against the misuse of genetic information, but they may not give full protection. There can also be a risk in knowing genetic information. There are laws against misuse of genetic information, but they may not give full protection. The Genetic Information Nondiscrimination Act of 2008, also referred to as GINA, was passed by Congress to protect Americans from such discrimination. The law prevents discrimination from health insurers and employers. This law does not cover life insurance, disability insurance and long-term care insurance. New health information about inherited traits that might affect you or your blood relatives could be found during a study. The researchers believe the chance these things will happen is very small, but cannot promise that they will not occur.

#### HOW WILL INFORMATION ABOUT ME BE KEPT PRIVATE?

Your privacy is very important to the researchers and they will make every effort to protect it. Here are just a few of the steps they will take:

- 1) When your samples are sent to the researchers, no information identifying you (such as your name) will be sent. Samples will be identified by a unique code only.
- 2) The list that links the unique code to your name will be kept separate from your sample and health information. Any Biobank and SWOG staff with access to the list must sign an agreement to keep your identity confidential.
- 3) Researchers to whom SWOG sends your sample and information will not know who you are. They must also sign an agreement that they will not try to find out who you are.
- 4) Information that identifies you will not be given to anyone, unless required by law.
- 5) If research results are published, your name and other personal information will not be used.

#### WHAT ARE THE POSSIBLE BENEFITS?

You will not benefit from taking part in this study.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

#### ARE THERE ANY COSTS OR PAYMENTS?

Neither you nor your health care plan/insurance carrier will be billed for the collection or testing of the tumor tissue or blood samples that will be used for this study. You will not be paid for taking part. If any of the research leads to new tests, drugs, or other commercial products, you will not share in any profits.



| WH | AT IF I CHANC | GE MY MIND? |
|---|---|---|
| • | • | ger want your samples to be used, you can call the study doctor, sert name of study doctor for main trial) at |
| let th | e researchers know. | (insert telephone number of study doctor for main trial) who will Then, any sample that remains in the bank will no longer be used. |
| Samp | | nation that have already been given to or used by researchers will not be |
| WH | AT IF I HAVE N | MORE QUESTIONS? |
| | , (ins | out the use of your samples for research, contact the study doctor, ert name of study doctor for main trial), at |
| (inse | rt telephone number | of study doctor for main trial). |
| Pleas | | TURE RESEARCH STUDIES: to show whether or not you would like to take part in each option questions): |
| 1. | have an optional | bonds to treatment on this study, and then gets worse, I agree to biopsy to collect a sample of tissue. I agree to have this tumor d information kept in a Biobank for use in future health research. |
| 2. | My blood sample<br>future health rese<br>YES | es and related information may be kept in a Biobank for use in earch. NO |
| This | is the end of the sect | tion about optional studies. |
| My | Signature Agree | ing to Take Part in the Main Study |
| my q | uestions have been a | form, or had it read to me. I have discussed it with the study doctor and answered. I will be given a signed copy of this form. I agree to take part additional studies where I circled 'yes'. |
| Partic | cipant's signature | <u> </u> |
| Date | of signature | |

